CLINICAL TRIAL: NCT05495607
Title: Dialysis With CARPEDIEM®: French Multicentric Experience in 25 Patients
Brief Title: Continous Renal Replacement Therapy With the CARPEDIEM® in a French National Cohort of 25 Neonates and Small Infants
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22-NEPHRO-01
Record Dates: First submitted 2022-08-04; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Sepsis; Kidney Diseases; Metabolic Disease; Twin to Twin Transfusion Syndrome; Cardiac Disease; Pulmonary Disease
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Sepsis; Kidney Diseases; Metabolic Diseases; Fetofetal Transfusion; Heart Diseases; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: We have included 25 neonates and small infants having received CARPEDIEM® machine in France in a multicentric experience
  Interventions: Device: CARPEDIEN

INTERVENTIONS:
Device: CARPEDIEN — Continuous renal replacement therapy

SUMMARY:
Historically, CKRT and hemodialysis were performed in small infants and newborns with devices developed for adults with high rates of complications and mortality.

We aim to retrospectively report the first multicenter French experience of CARPEDIEM® use and evaluate the efficacy, feasibility, outcomes, and technical considerations of this new device in a population of neonates and small infant. Compared to adult's device continuous renal replacement therapy with an adapted machine allowed successful blood purification without severe complications even in low birth weight neonates.

ELIGIBILITY:
Inclusion criteria:

* Children and neonates including premature and low birth weight neonates
* Have a diagnosis of acute kidney injury, end stage renal disease, metabolic disease, electrolyte abnormality
* Require renal replacement therapy

Exclusion Criteria:

-Renal replacement therapy with another device than Carpediem machine

Ages: 0 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population will be selected in a department of pediatric and neonatal unit intensive care and whom need a renal replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Survival | 3 years
Serum creatinine | 3 years
Serum potassium | 3 years
Blood urea nitrogen | 3 years
Ammonia levels | 3 years

SECONDARY OUTCOMES:
Ultrafiltration flow | 3 years
  the substitution range with the effluent volume in ml/kg/h ( compared to the KDIGO recommend of 25-35 ml/kg/h)
Blood flow | 3 years
  The range of blood flow in ml/kg/min ( compared to the recommend blood flow of 3-10 ml/kg/min).
Anticoagulation | 3 years
  The dose of continuous heparin anticoagulation in UI/Kg/h to prevent circuit clotting.
Number of sessions | 3 years
Time of treatments | 3 years
CKRT modality | 3 years
Vascular access | 3 years
  The localization of a vascular access ( intern jugular, subclavian, umbilical or femoral).
Priming circuit | 3 years
  The priming circuit ( normal salin, albumin, Isofundin or packed red blood cells).
Size of the circuit | 3 years
Death | 3 years
Clotting circuit and other dysfunction circuit | 3 years
  * Dysfunction circuit included cathether dysfunction, pressure dysfucntion and failure restitution
  * Complications of an extra corporel therapy including hypotension, thrombocytopenia and clotting circuit.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No